CLINICAL TRIAL: NCT03016494
Title: A Randomized, Open-label, Oral Dose, Crossover Study to Evaluate the Pharmacokinetics and Safety of Fixed-dose Combination of DWJ1386 Compared With Co-administration of DWC20155 and DWC20156 in Healthy Subjects
Brief Title: Safety and Pharmacokinetics Study of Fixed Dose Combination of DWJ1386 Compared With Co-administration of DWC20155 and DWC20156 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWJ1386001
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test/Reference Drug (Experimental): DWJ1386 Tab. followed by co-administration of DWC20155 and DWC20156 Tab.
  Interventions: Drug: Co-administration of DWC20155 and DWC20156; Drug: DWJ1386 Tab.
- Reference/Test Drug (Experimental): co-administration of DWC20155 and DWC20156 Tab. followed by DWJ1386 Tab.
  Interventions: Drug: Co-administration of DWC20155 and DWC20156; Drug: DWJ1386 Tab.

INTERVENTIONS:
Drug: Co-administration of DWC20155 and DWC20156
Drug: DWJ1386 Tab.

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics between co-administration and fixed dose combination of DWC20155 and DWC20156 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* BMI≥18.5 and ≤27.0 kg/m2
* No clinically significant findings
* Age 19-55 years at screening

Exclusion Criteria:

* Who has allergy to investigational product

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0-24 hours
Area under the plasma concentration versus time curve (AUC) | 0-24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Busan Paik Hospital, Busan, Busanjin-gu, South Korea

IPD SHARING:
Plan to Share IPD: No